CLINICAL TRIAL: NCT00404196
Title: LEO19123 Cream in the Treatment of Hand Eczema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEO19123-C22
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2007-08

CONDITIONS: Hand Eczema
MeSH Terms: interventions — calcipotriene

INTERVENTIONS:
Drug: Calcipotriol and LEO80122 (LEO19123 cream)

SUMMARY:
To compare the efficacy and safety of two different dose combinations of LEO19123 cream (calcipotriol and LEO80122) with LEO19123 cream vehicle for 3 weeks in the treatment of patients with hand eczema.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hand eczema with or without atopic etiology/background
* Investigator.s Global Assessment of disease severity graded as at least mild at Visit 1
* Patients should be Caucasian males aged from 18 years
* Attending a hospital outpatient clinic or the private practise of a dermatologist.
* Following verbal and written information about the trial, the patient must provide signed and dated informed consent before any trial related activity is carried out, including activities relating to wash-out periods.

Exclusion Criteria:

* Systemic treatment with immunosuppressive drugs (e.g. methotrexate, cyclosporine, azathioprine) or corticosteroids within 4 weeks prior to randomisation. (Inhaled or intranasal steroids for asthma or rhinitis may be used).
* PUVA or UVB therapy on the hands within 4 weeks prior to randomisation.
* Topical treatment with immunomodulators (pimecrolimus, tacrolimus) or corticosteroids from WHO groups III or IV on the hands within 2 weeks prior to randomisation.
* Other topical therapy on the hands (except for the use of emollient) within 1 week prior to randomisation.
* Use of other treatment (drug, non-drug) on the hands during the trial except for the use of investigational product and emollient.
* Concurrent skin diseases on the hands.
* Current diagnosis of exfoliative dermatitis.
* Significant clinical infection (impetiginised hand eczema) on the hands, which requires antibiotic treatment.
* Known or suspected hypersensitivity to component(s) of the investigational product.
* Positive patch test as defined in protocol
* Known or suspected severe renal insufficiency or severe hepatic disorders.
* Patients with history/signs/symptoms suggestive of an abnormality of calcium homeostasis associated with clinically significant hypercalcaemia.
* Patients with history of cancer except for basal cell carcinoma.
* Current participation in any other interventional clinical trial.
* Patients who have received treatment with any nonmarketed drug substance (i.e. an agent which has not yet been made available for clinical use following registration) within 4 weeks prior to randomisation.
* Previously randomised in this study.
* Patients known or, in the opinion of the investigator, is unlikely to comply with the Clinical Study Protocol (e.g. alcoholism, drug dependency, or psychotic state).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-10; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Proof of concept

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- Queen's Medical Centre, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No